CLINICAL TRIAL: NCT01841554
Title: Cardioband Adjustable Annuloplasty System For Transcatheter Repair of Mitral Valve Regurgitation
Brief Title: Cardioband With Transfemoral Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB1-1/CB1-2; NCT01533883 (obsolete NCT alias)
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Mitral Regurgitation
Keywords: Mitral Valve; Annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental)
  Interventions: Device: Cardioband

INTERVENTIONS:
Device: Cardioband
  Other Names: With Transfemoral delivery system

SUMMARY:
To evaluate the performance and safety of the Cardioband Adjustable Annuloplasty System for repair of functional mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Moderate to severe functional Mitral Regurgitation (MR)
* Symptomatic Patients (NYHA ClassII-IV) despite optimal medical therapy , including Cardiac Resynchronization (CRT) if indicated.
* Left Ventricle Ejection Fraction (LVEF) ≥ 25%, LVEDD ≤ 65mm
* Subject is high risk to undergo Mitral Valve (MV) surgery (as assessed by a surgeon and a cardiologist, at the site)
* Transseptal catheterization and femoral vein access is determined to be feasible
* Subject is able and willing to give informed consent and follow protocol procedures

Exclusion Criteria:

* Active bacterial endocarditis
* Severe organic lesions with retracted chordae or congenital malformations with lack of valvular tissue
* Heavily calcified annulus or leaflets
* Subjects in whom transesophageal echocardiography is contraindicated
* Untreated clinically significant Coronary Artery Disease (CAD) requiring revascularization
* CRT implant within 3 months prior to procedure
* Any percutaneous coronary, carotid, endovascular intervention or carotid surgery within 30 days or any coronary or endovascular surgery within 3 months
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) within 6 months or severe carotid stenosis (>70% by Ultra sound)
* Renal insufficiency requiring dialysis
* Life expectancy of less than twelve months
* Subject is participating in concomitant research studies of investigational products
* Mitral valve anatomy which may preclude proper device treatment
* Right-sided congestive heart failure with echocardiographic evidence of severe right ventricular dysfunction and severe tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maisano, Prof., Principal Investigator — Universitätsspital Zürich
Locations (11):
- Hôpital Bichat-Claude Bernard, Paris, France
- Germany (5):
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik II, Bonn
  - Universitätskliniken zu Köln Klinik III Innere Medizin, Cologne
  - Asklepios Klinik, St. Georg, Hamburg
  - Zentrum für Kardiologie, Universitätsmedizin Mainz, Mainz
  - Munich University Clinic, Munich
- Rambam Cardiology Research Unit, Haifa, Israel
- Italy (2):
  - Azienda Ospedaliero - Universitaria "Policlinico - Vittorio Emanuele", Catania
  - San Raffaele University Hospital, Milan
- St.Antonius Ziekenhuis, Nieuwegein, Netherlands
- UniversitätsSpital Zürich, Zurich, Switzerland

REFERENCES:
- [Background] Maisano F, La Canna G, Latib A, Denti P, Taramasso M, Kuck KH, Colombo A, Alfieri O, Guidotti A, Messika-Zeitoun D, Vahanian A. First-in-man transseptal implantation of a "surgical-like" mitral valve annuloplasty device for functional mitral regurgitation. JACC Cardiovasc Interv. 2014 Nov;7(11):1326-8. doi: 10.1016/j.jcin.2014.08.003. Epub 2014 Oct 15. No abstract available. PMID 25326746
- [Background] Maisano F, Taramasso M, Nickenig G, Hammerstingl C, Vahanian A, Messika-Zeitoun D, Baldus S, Huntgeburth M, Alfieri O, Colombo A, La Canna G, Agricola E, Zuber M, Tanner FC, Topilsky Y, Kreidel F, Kuck KH. Cardioband, a transcatheter surgical-like direct mitral valve annuloplasty system: early results of the feasibility trial. Eur Heart J. 2016 Mar 7;37(10):817-25. doi: 10.1093/eurheartj/ehv603. Epub 2015 Nov 18. PMID 26586779
- [Derived] Messika-Zeitoun D, Nickenig G, Latib A, Kuck KH, Baldus S, Schueler R, La Canna G, Agricola E, Kreidel F, Huntgeburth M, Zuber M, Verta P, Grayburn P, Vahanian A, Maisano F. Transcatheter mitral valve repair for functional mitral regurgitation using the Cardioband system: 1 year outcomes. Eur Heart J. 2019 Feb 1;40(5):466-472. doi: 10.1093/eurheartj/ehy424. PMID 30124798
- [Derived] Nickenig G, Hammerstingl C, Schueler R, Topilsky Y, Grayburn PA, Vahanian A, Messika-Zeitoun D, Urena Alcazar M, Baldus S, Volker R, Huntgeburth M, Alfieri O, Latib A, La Canna G, Agricola E, Colombo A, Kuck KH, Kreidel F, Frerker C, Tanner FC, Ben-Yehuda O, Maisano F. Transcatheter Mitral Annuloplasty in Chronic Functional Mitral Regurgitation: 6-Month Results With the Cardioband Percutaneous Mitral Repair System. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2039-2047. doi: 10.1016/j.jcin.2016.07.005. PMID 27712741

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 62 patients originally enrolled, 1 excluded from full analysis data set (N=61) but included in safety analysis data set (N=62). Patient had severe MR, right heart failure (RHF), and tricuspid regurgitation (TR); determined to be a significant deviation from intended use of device. Study protocol amended to exclude severe RHF and TR.
Groups:
- Single: Multi-center, prospective study with intra-subject comparisons
Period: Overall Study
Arm/Group | Single
Started | 61
Implanted | 60
1 Year Follow Up | 42
Completed | 42
Not Completed | 19
Not completed — Death | 7
Not completed — No Implantation | 1
Not completed — Discontinued Follow Up | 5
Not completed — Study exit due to secondary intervention | 6

BASELINE CHARACTERISTICS:
Arm/Group | Single
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 44
EuroSCORE II [Mean (Standard Deviation); unit: Score] — EuroScore II is a risk model which allows the calculation of the risk of death after a heart operation.
  EuroScore II risk levels are as follows:
  * < 8: Low risk
  * 8-10: Moderate risk
  * >10: High risk
  Score | 7.3 (6.3)
New York Heart Association (NYHA) Functional Class III or IV [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure:
  1. Class I - No symptoms and no limitation in ordinary physical activity
  2. Class II - Mild symptoms and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants | 52
Ischemic Etiology of Regurgitation [Count of Participants; unit: Participants] | 37
Left Ventricule Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percent Fraction] | 33 (11)
Previous Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] — Population: Data Unavailable for 2 patients.
  Participants
    number analyzed (Participants) | 59
    (all) | 18
Renal Insufficiency [Count of Participants; unit: Participants] | 49
Atrial Fibrillation [Count of Participants; unit: Participants] — Population: Data unavailable for 1 patient.
  Participants
    number analyzed (Participants) | 60
    (all) | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Serious Adverse Events and Serious Adverse Device Effects
Description: Overall rate of Major Serious Adverse Events (SAEs) and serious adverse device effects (SADEs) until hospital discharge and at post-operative 30 days.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 61
Participants
  Death | 2
  Myocardial Infarction | 1
  Major Bleeding Complications | 2
  Renal Failure | 4
  Cardiac Tamponade | 1
  Respiratory Failure | 0

2. Secondary Outcome: Performance [6MWT]
Description: Distance in meters walked during 6 Minute Walk Test (6MWT) at baseline, 6 and 12 months.
Time Frame: Baseline, 6 and 12 months
Population: Intra-subject comparison of 18 patients who had data at all three time points (baseline, 6 and 12 months).
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Single
Number analyzed (Participants) | 18
Meters
  Baseline | 334.7778 (120.3957)
  6 Months | 393.2222 (114.4529)
  1 Year | 407.0556 (122.8899)

3. Secondary Outcome: Performance [MLHFQ]
Description: Score on Minnesota Living with Heart Failure Questionnaire (MLHFQ). MLHFQ is composed of 21 questions relating to limitations in lifestyle associated with heart failure. Respondents use a 5 point scale from 0 to 5, with a 0 representing no limitation and 5 representing maximum limitation. The total score is computed by adding individual scores of each question. Higher scores are associated with lower quality of life.
Time Frame: Baseline, 6 and 12 months
Population: Intra-subject comparison of 27 patients who had data at all three time points (baseline, 6 and 12 months).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single
Number analyzed (Participants) | 27
Scores on a scale
  Baseline | 35.8889 (16.6579)
  6 Months | 16.2593 (14.9244)
  1 Year | 19.3333 (19.9538)

4. Secondary Outcome: Performance [Intra-subject Comparison - MR Severity]
Description: All data available at each time point was reported as number of patients with MR grades between 0-1 (Trace - Mild), 2+ (Moderate), 3-4+ (Moderate - Severe).
Time Frame: Baseline, discharge, 6 and 12 months
Population: Intra-subject comparison of 26 patients who were assessed for MR grade across all four time points (baseline, discharge, 6 and 12 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 26
Participants
  Baseline: Moderate - Severe (3-4+) | 16
  Baseline: Moderate (2+) | 10
  Baseline: Trace - Mild (0-1+) | 0
  Discharge: Moderate - Severe (3-4+) | 1
  Discharge: Moderate (2+) | 5
  Discharge: Trace - Mild (0-1+) | 20
  6 Months: Moderate - Severe (3-4+) | 0
  6 Months: Moderate (2+) | 5
  6 Months: Trace - Mild (0-1+) | 21
  1 Year: Moderate - Severe (3-4+) | 0
  1 Year: Moderate (2+) | 7
  1 Year: Trace - Mild (0-1+) | 19

5. Secondary Outcome: Performance [Full Analysis Data Set - MR Severity]
Description: as for outcome 4
Time Frame: Baseline, discharge, 6 and 12 months
Population: The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 61
Participants
  Baseline: Moderate - Severe (3-4+) | 45
  Baseline: Moderate (2+) | 16
  Baseline: Trace - Mild (0-1+) | 0
  Discharge: number analyzed (Participants) | 58
  Discharge: Moderate - Severe (3-4+) | 6
  Discharge: Moderate (2+) | 13
  Discharge: Trace - Mild (0-1+) | 39
  6 Months: number analyzed (Participants) | 43
  6 Months: Moderate - Severe (3-4+) | 3
  6 Months: Moderate (2+) | 11
  6 Months: Trace - Mild (0-1+) | 29
  1 Year: number analyzed (Participants) | 39
  1 Year: Moderate - Severe (3-4+) | 2
  1 Year: Moderate (2+) | 10
  1 Year: Trace - Mild (0-1+) | 27

6. Other Pre Specified Outcome: Reduce MR [Paired Baseline and Follow-Up]
Description: Cardioband ability to reduce mitral valve regurgitation (MR) Intra-procedure, at hospital discharge, and at 30 days. Reported as number of patients showing a reduction in MR grade greater than or equal to 1.
Time Frame: Post-adjustment, discharge, and 30 Days
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and post-adjustment, discharge, and 30 days is 47, 50 and 46, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 58
Participants
  Post-Adjustment: number analyzed (Participants) | 52
  Post-Adjustment | 47
  Discharge | 50
  30 Days: number analyzed (Participants) | 54
  30 Days | 46

7. Other Pre Specified Outcome: Technical Feasibility of Cardioband Adjustment
Description: The ability to connect the Adjustment Tool, reduce septo-lateral dimension, and retract the Adjustment Tool with guide wire.
Time Frame: Immediately after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 61
Participants | 58

8. Other Pre Specified Outcome: Technical Success Rate of the Implantation of the Cardioband
Description: The ability to advance the implant, load anchors, anchor the implant to tissue, and retract the Implant Delivery System.
Time Frame: Immediately after implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 61
Participants | 60

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Of 62 patients originally enrolled in the study, one had severe MR, severe right heart failure (RHF), and severe tricuspid regurgitation (TR). The CEC determined this was a significant deviation from the intended use of the device. The study protocol was amended to exclude severe RHF and severe TR to emphasize this patient's condition did not fit the intended use of the device. The patient was excluded from the full analysis data set (N=61) but included in the safety analysis data set (N=62).
Arm/Group | Single
Serious Adverse Events (participants affected / at risk) | 44/62
Other Adverse Events (participants affected / at risk) | 21/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=62)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) — CEC Adjudicated
Atrial Fibrillation (Cardiac disorders) | 2 (2) — CEC Adjudicated
Atrial Septal Defect (Cardiac disorders) | 1 (1) — CEC Adjudicated
Bundle Branch Block Left (Cardiac disorders) | 2 (2) — CEC Adjudicated
Cardiac Arrest (Cardiac disorders) | 2 (2) — CEC Adjudicated
Cardiac Failure (Cardiac disorders) | 15 (22) — CEC Adjudicated
Cardiac Tamponade (Cardiac disorders) | 1 (1) — CEC Adjudicated
Cardiogenic Shock (Cardiac disorders) | 1 (1) — CEC Adjudicated
Dyspnoea (Cardiac disorders) | 1 (1) — CEC Adjudicated
Left Ventricular Failure (Cardiac disorders) | 1 (1) — CEC Adjudicated
Mitral Valve Disease (Cardiac disorders) | 4 (4) — CEC Adjudicated
Myocardial Infarction (Cardiac disorders) | 2 (3) — CEC Adjudicated
Pericardial Effusion (Cardiac disorders) | 3 (4) — CEC Adjudicated
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) — CEC Adjudicated
Ventricular Tachycardia (Cardiac disorders) | 3 (3) — CEC Adjudicated
Cataract (Eye disorders) | 1 (1) — CEC Adjudicated
Melaena (Gastrointestinal disorders) | 1 (1) — CEC Adjudicated
Chest Pain (General disorders) | 1 (1) — CEC Adjudicated
Device Dislocation (General disorders) | 1 (1) — CEC Adjudicated
Multi-Organ Failure (General disorders) | 1 (1) — CEC Adjudicated
Oedema due to Cardiac Disease (General disorders) | 2 (2) — CEC Adjudicated
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) — CEC Adjudicated
Pneumonia (Infections and infestations) | 2 (2) — CEC Adjudicated
Sepsis (Infections and infestations) | 1 (1) — CEC Adjudicated
Septic Shock (Infections and infestations) | 2 (2) — CEC Adjudicated
Staphylococcal Infection (Infections and infestations) | 1 (1) — CEC Adjudicated
Urinary Tract Infection (Infections and infestations) | 1 (1) — CEC Adjudicated
Contusion (Injury, poisoning and procedural complications) | 1 (1) — CEC Adjudicated
Iatrogenic Injury (Injury, poisoning and procedural complications) | 2 (2) — CEC Adjudicated
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — CEC Adjudicated
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — CEC Adjudicated
Blood Glucose Increased (Investigations) | 1 (2) — CEC Adjudicated
Haemoglobin Decreased (Investigations) | 1 (1) — CEC Adjudicated
Troponin Increased (Investigations) | 1 (1) — CEC Adjudicated
Dehydration (Metabolism and nutrition disorders) | 1 (1) — CEC Adjudicated
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (2) — CEC Adjudicated
Meniscus Injury (Musculoskeletal and connective tissue disorders) | 1 (1) — CEC Adjudicated
Carcinoma in situ of Eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — CEC Adjudicated
Large Intestine Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) — CEC Adjudicated
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — CEC Adjudicated
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) — CEC Adjudicated
Hemiparesis (Nervous system disorders) | 1 (1) — CEC Adjudicated
Ischaemic Stroke (Nervous system disorders) | 1 (1) — CEC Adjudicated
Syncope (Nervous system disorders) | 1 (1) — CEC Adjudicated
Renal Failure (Renal and urinary disorders) | 4 (8) — CEC Adjudicated
Actinomycotic Pulmonary Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — CEC Adjudicated
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — CEC Adjudicated
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — CEC Adjudicated
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — CEC Adjudicated
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) — CEC Adjudicated
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1) — CEC Adjudicated
Hospitalisation (Surgical and medical procedures) | 1 (1) — CEC Adjudicated
Implantable Defibrillator Insertion (Surgical and medical procedures) | 1 (1) — CEC Adjudicated
Air Embolism (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=62)
Atrial Fibrillation (Cardiac disorders) | 6 (6)
Device Fastener Issue (General disorders) | 4 (4)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Haemoglobin Decreased (Investigations) | 4 (4)
Renal Failure (Renal and urinary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes